CLINICAL TRIAL: NCT04726462
Title: Comparison of the Effects of Two Different Exercise Programs on Lower Extremity Functions, Posture and Physical Activity in Office Workers
Brief Title: Comparison of the Effects of Two Different Exercise Programs in Office Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nilay Arman, Assist. Prof., Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12259
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Physical Activity; Exercise; Office Worker; Lower Extremity Function; Posture
Keywords: Physical Activity; Exercise; Office Worker; Lower Extremity Function; Posture
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional exercise group (Experimental)
  Interventions: Other: Functional exercises
- Posture exercises group (Experimental)
  Interventions: Other: Posture exercises

INTERVENTIONS:
Other: Functional exercises — The exercise program is planned as a function-oriented exercise program aimed at improving balance skills, increasing lower extremity muscle strength and functions.
  Arms: Functional exercise group
Other: Posture exercises — The exercise program was planned by focusing on posture exercises in order to increase the postural smoothness of the participants.
  Arms: Posture exercises group

SUMMARY:
The aim of our study is to compare the effects of functional exercises and posture exercises on lower extremity functions, posture and physical activity in office workers. For this reason, functional exercises will be applied to a group of office workers and posture exercises will be applied to a group, lower extremity functions, posture and physical activity will be evaluated before and after the training.

DETAILED DESCRIPTION:
There are studies reporting that the long working time spent at the desk in office workers and working in a static position are the etiological factors of various problems in the upper and lower extremities.Office workers who are eligible for inclusion criteria and willing to participate in the study will be included.Participants will be randomly divided into two groups as functional exercise group and posture exercises group.

Exercise program:

1. st Group: Functional exercise group (20 people) The exercise program is planned as a function-oriented exercise program aimed at improving balance skills, increasing lower extremity muscle strength and functions. During all exercises, exercises will be done while maintaining postural smoothness. For the postural smoothness, feedback will be provided by the physiotherapist for orientation, correction and protection to the participants. The exercise program will be applied online, 2 days a week for 8 weeks. In the beginning, 3 sets of 10 repetitions will be progressed gradually as 3 sets of 15 repetitions, 3 sets of 20 repetitions, according to the tolerance of the participant. Exercises will be progressed from simple to difficult. There will be a 2-minute rest period between sets. All 28 exercises defined in the functional exercise group will not be applied in one session. Exercise selection will be made according to the functional status of the participant.Exercises are planned to be performed in a chair supported, bipedal position, unipedal position, using weights, providing resistance with elastic band in various degrees of difficulty and in various positions. In the beginning, 6-7 exercises, which are appropriate according to the evaluation results of the participants, will be selected according to the difficulty level and the exercises will be changed in the following weeks. The exercises will start with warm-up exercises and end with cooling exercises. Warm-up exercises and cool-down exercises will take 5 minutes at the beginning and 5 minutes at the end, a total of 10 minutes.
2. nd Group: Posture exercises group (20 people) The exercise program was planned by focusing on posture exercises in order to increase the postural smoothness of the participants. During all exercises, exercises will be done while maintaining postural smoothness. For the postural smoothness, feedback will be provided by the physiotherapist for orientation, correction and protection to the participants. The exercise program will be applied online, 2 days a week for 8 weeks. In the beginning, range of motion exercises will be progressed as 3 sets of 10 repetitions, then gradually as 3 sets of 15 repetitions and 3 sets of 20 repetitions, according to the tolerance of the participant. Stretching exercises will be done as 3 sets of 6-8 repetitions. Initially, 6-7 exercises will be selected according to the postural evaluation results of the participants.

Exercises will be changed in the following weeks. Resistance will not be applied in the exercises, and the participants will be asked to maintain the specified exercise position for 5-6 seconds for range of motion exercises and 20 30 seconds for stretching exercises.

ELIGIBILITY:
Inclusion Criteria:

* Being in the age range of 20-45
* Being an office worker Working remotely and alternately due to the Covid 19 pandemic
* Working at the computer for at least 4-5 hours a day

Exclusion Criteria:

* Having a surgical history of the lower extremity Presence of a chronic neurological, orthopedic, vestibular or cardiac disease
* Being pregnant
* Exercising regularly or doing sports for the past year

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
6 Minute Walking Test (6 MWT) | Change from baseline to 8 weeks, follow up at two months
  The six-minute walk test is an example of a timed distance test that is widely used in clinical research and rehabilitation studies. It can be applied in a short time. Requires little equipment. Used as a field test, the six minute walk test is a simple and straightforward walk test that does not need exercise equipment, compatible with daily activities it is an inexpensive test. Before the test begins, the patient is seated in a chair near the starting point for at least 10 minutes should rest. The walking area should be at least 30 m long. A shorter corridor is more for more frequent turns and changes of direction. It takes a lot of time. It is kept for 6 minutes with the help of the stopwatch and the number of laps in the time is calculated and saved. 6 MWTs will be used to evaluate the lower extremity functions of the cases included in the study.
Sit to Stand Test | Change from baseline to 8 weeks, follow up at two months
  It reflects lower extremity muscle strength and functional capacities of individuals. For the test, the individual is allowed to sit in the middle of a chair with a height of 43.18 cm, with his back upright, with his feet on the ground and arms crossed in front of his chest (right hand left shoulder, left hand on the right shoulder). While the individual is in this position, the test starts with the start command and the total number of starts made during 30 seconds creates the individual's score. One of the aims of our study is to investigate the effects of exercise programs on lower extremity functions of office workers. For this reason, sit and stand test will be used to evaluate lower extremity muscle strength for lower extremity functions of the cases included in the study.
10 Step Up Time Test | Change from baseline to 8 weeks, follow up at two months
  All cases are asked to climb 10 steps (14x28x120 cm) as fast as possible. Step-up time is measured by the stopwatch in seconds. The measurement is repeated three times and the average of the three measurements is recorded. One of the aims of our study is to investigate the effects of exercise programs on lower extremity functions of office workers. For this reason, the 10-step climbing time test will be used to evaluate the lower extremity functions of the cases included in the study.
PostureScreen Mobile | Change from baseline to 8 weeks, follow up at two months
  There are different systems that use digital photographs and software analysis to evaluate posture. PostureScreen Mobile (posture analysis / body composition / motion evaluation software) is a valid and reliable application developed to evaluate posture with the help of a camera system.
International physical activity questionnaire-short form | Change from baseline to 8 weeks, follow up at two months
  In the survey, the time that individuals have physically spent in the last 7 days and the types of physical activity they do in their daily lives questioned by considering
Functional Reach Test | Change from baseline to 8 weeks, follow up at two months
  This test evaluates postural stability by measuring the maximum stretched distance.
Semi-squat test | Change from baseline to 8 weeks, follow up at two months
  Participants are asked to stay in a half-squatting position on a hard surface, without shoes, with feet shoulder-width apart, arms crossed on the chest and the body upright.

CONTACTS AND LOCATIONS:
Locations (1):
- Aysenur Namli, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Namli Seker A, Arman N. Comparison of the Effects of Two Different Exercise Programs on Lower Limb Functions, Posture, and Physical Activity in Office Workers Working at Home and in Office Alternately: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2024 Feb 1;103(2):134-142. doi: 10.1097/PHM.0000000000002315. Epub 2023 Jul 18. PMID 37535624